CLINICAL TRIAL: NCT02373774
Title: Sonographic Visualization vs Palpation Technique for Infant Lumbar Puncture
Brief Title: Ultrasound vs Palpation for Infant Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, David Kessler, Assistant Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AAAO3705
Record Dates: First submitted 2015-02-07; First posted 2015-02-27 (Estimated); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Spinal; Puncture, Complications
Keywords: infant; lumbar puncture; patient safety; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Anatomic Palpation Technique (No Intervention): Participants randomized to this group will receive standard of care treatment with providers using the palpation technique to select an interspace to perform lumbar puncture.
- Pre-Procedural Ultrasound (Experimental): Participants randomized to this group will receive an ultrasound of the interspace selected via the palpation method prior to performance of the lumbar puncture to determine measurements of appropriate angle and depth and evaluation of any overlying vasculature.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Patients will receive an ultrasound prior to lumbar puncture procedure to help visualize and select spinal interspace.
  Other Names: (Zonare Z1.pro and/or Sonosite Mturbo)
  Arms: Pre-Procedural Ultrasound

SUMMARY:
The purpose of this study is to determine if performing an ultrasound to identify the space to insert the needle before performing a lumbar puncture will improve success of the procedure and patient safety.

DETAILED DESCRIPTION:
The investigators are conducting a single-center, prospective two-arm parallel group randomized clinical trial in an urban pediatric emergency department to determine if performing an ultrasound prior to lumbar puncture procedure improves success of the procedure.

Patients will be block-randomized into two groups to receive procedural interspace selection via 1) standard anatomic palpation technique or 2) visualization with pre-procedural ultrasound (experimental group).

1. Standard Anatomic Palpation Technique:

   Participants randomized to this group will receive standard of care treatment with providers using the palpation technique to select an interspace. As variations on the palpation technique exist, the investigators will provide a standardized educational cognitive aid that clinicians can use for this approach.
2. Pre-Procedural Ultrasound:

Clinicians will first use the standard palpation technique to select an interspace for ultrasound evaluation. A select group of pediatric emergency medicine attendings and fellows who have already trained to a mastery standard with the ultrasound protocol will then conduct the pre-procedural ultrasound. The clinicians performing the lumbar puncture will be provided the following information to conduct the lumbar puncture:

i. Assessment for fluid at the level selected (and the number of interspaces above that have fluid without conus present)

ii. Measurements of appropriate angle and depth

iii. Evaluation of any overlying vasculature

Post-Lumbar Puncture:

After the lumbar puncture, infants randomized to both groups will receive a post-procedural ultrasound scan performed by one of the mastery trained ultrasound physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient is less than 90 days old.
* Patient is receiving a lumbar puncture

Exclusion Criteria:

* Patient is clinically unstable
* Patient had a previous lumbar puncture in the past 24 hours
* An outside consultant (not working in ED) is performing the LP
* Patient has developmental delay or neurological impairment
* There is no legal guardian present
* The legal guardians speak neither English nor Spanish
* There is no ultrasound personnel available to enroll

Max Age: 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O Kessler, MD, MSc, Principal Investigator — Columbia University; Gerald Behr, MD, Principal Investigator — Columbia University; Peter S Dayan, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Alpern ER, Stanley RM, Gorelick MH, Donaldson A, Knight S, Teach SJ, Singh T, Mahajan P, Goepp JG, Kuppermann N, Dean JM, Chamberlain JM; Pediatric Emergency Care Applied Research Network. Epidemiology of a pediatric emergency medicine research network: the PECARN Core Data Project. Pediatr Emerg Care. 2006 Oct;22(10):689-99. doi: 10.1097/01.pec.0000236830.39194.c0. PMID 17047467
- [Background] Jain S, Cheng J, Alpern ER, Thurm C, Schroeder L, Black K, Ellison AM, Stone K, Alessandrini EA. Management of febrile neonates in US pediatric emergency departments. Pediatrics. 2014 Feb;133(2):187-95. doi: 10.1542/peds.2013-1820. Epub 2014 Jan 27. PMID 24470644
- [Background] Kessler DO, Arteaga G, Ching K, Haubner L, Kamdar G, Krantz A, Lindower J, Miller M, Petrescu M, Pusic MV, Rocker J, Shah N, Strother C, Tilt L, Weinberg ER, Chang TP, Fein DM, Auerbach M. Interns' success with clinical procedures in infants after simulation training. Pediatrics. 2013 Mar;131(3):e811-20. doi: 10.1542/peds.2012-0607. Epub 2013 Feb 25. PMID 23439901
- [Background] Nigrovic LE, Kuppermann N, Neuman MI. Risk factors for traumatic or unsuccessful lumbar punctures in children. Ann Emerg Med. 2007 Jun;49(6):762-71. doi: 10.1016/j.annemergmed.2006.10.018. Epub 2007 Feb 23. PMID 17321005
- [Background] Glatstein MM, Zucker-Toledano M, Arik A, Scolnik D, Oren A, Reif S. Incidence of traumatic lumbar puncture: experience of a large, tertiary care pediatric hospital. Clin Pediatr (Phila). 2011 Nov;50(11):1005-9. doi: 10.1177/0009922811410309. Epub 2011 May 27. PMID 21622691
- [Background] Bonadio W. Pediatric lumbar puncture and cerebrospinal fluid analysis. J Emerg Med. 2014 Jan;46(1):141-50. doi: 10.1016/j.jemermed.2013.08.056. Epub 2013 Nov 1. PMID 24188604
- [Background] Duniec L, Nowakowski P, Kosson D, Lazowski T. Anatomical landmarks based assessment of intravertebral space level for lumbar puncture is misleading in more than 30%. Anaesthesiol Intensive Ther. 2013 Jan-Mar;45(1):1-6. doi: 10.5603/AIT.2013.0001. PMID 23572300
- [Background] Furness G, Reilly MP, Kuchi S. An evaluation of ultrasound imaging for identification of lumbar intervertebral level. Anaesthesia. 2002 Mar;57(3):277-80. doi: 10.1046/j.1365-2044.2002.2403_4.x. PMID 11892638
- [Background] Shekelle PG, Wachter RM, Pronovost PJ, Schoelles K, McDonald KM, Dy SM, Shojania K, Reston J, Berger Z, Johnsen B, Larkin JW, Lucas S, Martinez K, Motala A, Newberry SJ, Noble M, Pfoh E, Ranji SR, Rennke S, Schmidt E, Shanman R, Sullivan N, Sun F, Tipton K, Treadwell JR, Tsou A, Vaiana ME, Weaver SJ, Wilson R, Winters BD. Making health care safer II: an updated critical analysis of the evidence for patient safety practices. Evid Rep Technol Assess (Full Rep). 2013 Mar;(211):1-945. PMID 24423049
- [Background] Coley BD, Shiels WE 2nd, Hogan MJ. Diagnostic and interventional ultrasonography in neonatal and infant lumbar puncture. Pediatr Radiol. 2001 Jun;31(6):399-402. doi: 10.1007/s002470100453. PMID 11436885
- [Background] Abo A, Chen L, Johnston P, Santucci K. Positioning for lumbar puncture in children evaluated by bedside ultrasound. Pediatrics. 2010 May;125(5):e1149-53. doi: 10.1542/peds.2009-0646. Epub 2010 Apr 19. PMID 20403933
- [Background] Lo MD, Parisi MT, Brown JC, Klein EJ. Sitting or tilt position for infant lumbar puncture does not increase ultrasound measurements of lumbar subarachnoid space width. Pediatr Emerg Care. 2013 May;29(5):588-91. doi: 10.1097/PEC.0b013e31828e630d. PMID 23603648
- [Background] Oncel S, Gunlemez A, Anik Y, Alvur M. Positioning of infants in the neonatal intensive care unit for lumbar puncture as determined by bedside ultrasonography. Arch Dis Child Fetal Neonatal Ed. 2013 Mar;98(2):F133-5. doi: 10.1136/archdischild-2011-301475. Epub 2012 Jun 9. PMID 22684159
- [Background] Shaikh F, Brzezinski J, Alexander S, Arzola C, Carvalho JC, Beyene J, Sung L. Ultrasound imaging for lumbar punctures and epidural catheterisations: systematic review and meta-analysis. BMJ. 2013 Mar 26;346:f1720. doi: 10.1136/bmj.f1720. PMID 23532866
- [Background] Bruccoleri RE, Chen L. Needle-entry angle for lumbar puncture in children as determined by using ultrasonography. Pediatrics. 2011 Apr;127(4):e921-6. doi: 10.1542/peds.2010-2511. Epub 2011 Mar 28. PMID 21444601
- [Background] Bailie HC, Arthurs OJ, Murray MJ, Kelsall AW. Weight-based determination of spinal canal depth for paediatric lumbar punctures. Arch Dis Child. 2013 Nov;98(11):877-80. doi: 10.1136/archdischild-2013-303793. Epub 2013 Aug 21. PMID 23966025
- [Background] Wilson DA, Prince JR. John Caffey award. MR imaging determination of the location of the normal conus medullaris throughout childhood. AJR Am J Roentgenol. 1989 May;152(5):1029-32. doi: 10.2214/ajr.152.5.1029. PMID 2650477
- [Background] Hill CA, Gibson PJ. Ultrasound determination of the normal location of the conus medullaris in neonates. AJNR Am J Neuroradiol. 1995 Mar;16(3):469-72. PMID 7793365
- [Background] Wolf S, Schneble F, Troger J. The conus medullaris: time of ascendence to normal level. Pediatr Radiol. 1992;22(8):590-2. doi: 10.1007/BF02015359. PMID 1491937
- [Background] Sahin F, Selcuki M, Ecin N, Zenciroglu A, Unlu A, Yilmaz F, Mavis N, Saribas S. Level of conus medullaris in term and preterm neonates. Arch Dis Child Fetal Neonatal Ed. 1997 Jul;77(1):F67-9. doi: 10.1136/fn.77.1.f67. PMID 9279188
- [Background] Rozzelle CJ, Reed GT, Kirkman JL, Shannon CN, Chern JJ, Wellons JC 3rd, Tubbs RS. Sonographic determination of normal Conus Medullaris level and ascent in early infancy. Childs Nerv Syst. 2014 Apr;30(4):655-8. doi: 10.1007/s00381-013-2310-6. Epub 2013 Nov 1. PMID 24178234
- [Background] Tame SJ, Burstal R. Investigation of the radiological relationship between iliac crests, conus medullaris and vertebral level in children. Paediatr Anaesth. 2003 Oct;13(8):676-80. doi: 10.1046/j.1460-9592.2003.01120.x. PMID 14535904
- [Background] Kesler H, Dias MS, Kalapos P. Termination of the normal conus medullaris in children: a whole-spine magnetic resonance imaging study. Neurosurg Focus. 2007;23(2):E7. doi: 10.3171/FOC-07/08/E7. PMID 17961006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Anatomic Palpation Technique | Pre-Procedural Ultrasound
Started | 40 | 41
Completed | 40 | 38
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Anatomic Palpation Technique | Pre-Procedural Ultrasound | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 41 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 25.4 (19.4) | 29.9 (19.3) | 27.6 (NA) — The standard deviation for the entire group was not calculated at the time of data analysis. The standard deviation cannot be calculated without the raw data. The raw data have been destroyed as the study data retention period has passed. In addition, the study closed with the Institutional Review Board (IRB) in 2017 and further analysis cannot be conducted.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participant sex was not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Puncture Success - Composite Score Including Lab Results and Reported Attempts
Description: Our primary outcome of the clinical trial is binary, success or failure of lumbar puncture. Success is defined as obtaining a sample of cerebrospinal fluid on the first attempt that has a red blood cell count of <1000 red blood cells per high-powered field.
Time Frame: Outcome measured on the same day of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Anatomic Palpation Technique | Pre-Procedural Ultrasound
Number analyzed (Participants) | 40 | 38
Participants | 18 | 19

2. Secondary Outcome: Number of Attempts- Per Direct Observation
Description: Defined as the number of times a lumbar puncture needle is removed from skin and reinserted or a new needle is inserted.
Time Frame: Outcome measured at the time of the procedure (same day)
Measure: Median (Inter-Quartile Range); unit: number of attempts
Arm/Group | Standard Anatomic Palpation Technique | Pre-Procedural Ultrasound
Number analyzed (Participants) | 40 | 38
number of attempts | 2 [1 to 3] | 2 [1 to 2]

ADVERSE EVENTS:
Arm/Group | Standard Anatomic Palpation Technique | Pre-Procedural Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes